CLINICAL TRIAL: NCT03003598
Title: The Effects of Endotracheal Intubation Via McGrath Videolaryngoscope on Intraocular Pressure
Brief Title: The Effects of Intubation Via McGrath Videolaryngoscope on Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Selim Ozkan, M.D., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Asozkan-3
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Intraocular Pressure
Keywords: Intraocular pressure; videolaryngoscope; direct laryngoscope

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videolaryngoscopy (Active Comparator): Evaluate the difference between the two groups about hemodynamic and intraocular pressure responses.
  Interventions: Other: Videolaryngoscope
- Direct laryngoscopy (Active Comparator): Evaluate the difference between the two groups about hemodynamic and intraocular pressure responses.
  Interventions: Other: Direct laryngoscope

INTERVENTIONS:
Other: Videolaryngoscope — This device is used in endotracheal intubation and tonopen device for measuring of intraocular pressure. The investigators want to evaluate which one is better.
  Arms: Videolaryngoscopy
Other: Direct laryngoscope — This device is used in endotracheal intubation and tonopen device for measuring of intraocular pressure. The investigators want to evaluate which one is better.
  Arms: Direct laryngoscopy

SUMMARY:
In this study, the investigators aimed to compare the effects of endotracheal intubation via direct laryngoscope (DLS) and McGrath Videolaryngoscope (VL) on intraocular pressure.

DETAILED DESCRIPTION:
Total of 50 American Society of Anesthesiologist Grade 1-2, Mallampati score 1 or 2, age between 18 to 65 patient planned to undergo nonopthalmic surgery will be included to study. Patients with glaucoma, diabetes mellitus, cardiovascular and pulmonary diseases, American Society of Anesthesiologist Grade III and IV, Body mass index more than 35, difficult intubation, undergo obstetrical surgery and propofol, fentanyl, rocuronium contraindicated will be excluded from the study. Patients will be divided randomly into 2 groups as direct laryngoscopic and videolaryngoscopic intubation group. Patients will be preoxygenated with %100 O2 for 3 minutes then anesthesia will be induced using propofol 2 mg / kg, fentanyl 1 mcg/kg, and rocuronium 0,5 mg / kg in both groups. After 3 minutes mask ventilation, patients will be intubated (women with No:7-7,5, men with No:8-8,5 intubation tube) by oral route. systolic blood pressure, diastolic blood pressure, mean arterial pressure, peripheral oxygen saturation, perfusion indexwill be recorded and intraocular pressure measured by ophthalmologist by tonopen device will be recorded pre-induction (basal), after induction, 1,2,3,5 minutes after intubation, respectively. Period between handling of laryngoscope or videolaryngoscope after termination of mask ventilation and obtain end tidal carbon dioxide will be accepted as application time and recorded. Study will be terminated after 5th minute values taken.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologist) Grade 1-2,
* Mallampati score 1 or 2,
* Age between 18 to 65,
* Patient planned to undergo nonopthalmic surgery

Exclusion Criteria:

* Patients with glaucoma, diabetes mellitus, cardiovascular and pulmonary diseases, ASA Grade III and IV, BMI more than 35,
* Patients with difficult intubation,
* Patients undergoing obstetrical surgery and propofol, fentanyl, rocuronium contraindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | From Beginning of Anesthesia induction to 5th minutes of intubation
Heart rate | From Beginning of Anesthesia induction to 5th minutes of intubation
Intraocular pressure | From Beginning of Anesthesia induction to 5th minutes of intubation
Adverse events | within the first 24 hour after surgery

IPD SHARING:
Plan to Share IPD: Undecided